CLINICAL TRIAL: NCT03058237
Title: A Phase 1 Bioavailability Study of Arbaclofen Placarbil Modified Release Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: INDV-AP-102; 2016-003792-22 (EudraCT Number)
Record Dates: First submitted 2017-02-09; First posted 2017-02-20 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: The Clinical Trial Authorisation application for this study describes a flexible protocol design using the formulation design space concept to allow decision-making in response to interim PK observations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part 1: Regimen A (Experimental): One low dose Arbaclofen Placarbil MR Prototype A tablet taken under fasting conditions.
  Part 1 participants receive Regimens A, B, C, D and E in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A
- Part 1: Regimen B (Experimental): One low dose Arbaclofen Placarbil MR Prototype B tablet taken under fasting conditions.
  Part 1 participants receive Regimens A, B, C, D and E in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype B
- Part 1: Regimen C (Active Comparator): One low dose Arbaclofen Placarbil SR tablet taken under fasting conditions as the reference product.
  Part 1 participants receive Regimens A, B, C, D and E in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil SR
- Part 1: Regimen D (Experimental): One low dose tablet of the selected Arbaclofen Placarbil MR Prototype administered with 0.6 g/kg of beverage in orange juice.
  Part 1 participants receive Regimens A, B, C, D and E in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A; Drug: Arbaclofen Placarbil MR Prototype B
- Part 1: Regimen E (Experimental): An optional regimen of one low dose tablet of the selected Arbaclofen Placarbil MR Prototype administered with 0.6 g/kg of beverage in orange juice.
  Part 1 participants receive Regimens A, B, C, D and E in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A; Drug: Arbaclofen Placarbil MR Prototype B
- Part 2: Regimen F (Experimental): One low dose Arbaclofen Placarbil MR prototype tablet (selected based on review of the data in Part 1) taken under fasting conditions.
  Part 2 participants receive Regimens F, G, H, I and J in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A; Drug: Arbaclofen Placarbil MR Prototype B
- Part 2: Regimen G (Active Comparator): One low dose Arbaclofen Placarbil IR capsule taken under fasting conditions as the reference product.
  Part 2 participants receive Regimens F, G, H, I and J in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil IR
- Part 2: Regimen H (Experimental): One low dose Arbaclofen Placarbil MR prototype tablet (selected based on review of the data in Part 1) taken under fasting conditions.
  Part 2 participants receive Regimens F, G, H, I and J in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A; Drug: Arbaclofen Placarbil MR Prototype B
- Part 2: Regimen I (Experimental): One low dose Arbaclofen Placarbil MR prototype tablet (selected based on review of the data in Part 1) taken under fasting conditions.
  Part 2 participants receive Regimens F, G, H, I and J in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A; Drug: Arbaclofen Placarbil MR Prototype B
- Part 2: Regimen J (Experimental): One low dose Arbaclofen Placarbil MR prototype tablet (selected based on review of the data in Part 1) taken under fasting conditions, or a previously dosed MR prototype in the fed state. Part 2 participants receive Regimens F, G, H, I and J in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A; Drug: Arbaclofen Placarbil MR Prototype B
- Part 3: Regimen K (Experimental): One low dose selected Arbaclofen Placarbil MR prototype tablet (selected based on review of the data in Part 2) taken under fasting conditions.
  Part 3 participants receive Regimens K and L in a randomised crossover manner as the first two treatments, followed by Regimens M and N in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A; Drug: Arbaclofen Placarbil MR Prototype B
- Part 3: Regimen L (Experimental): One low dose selected Arbaclofen Placarbil MR prototype tablet administered with 0.6 g/kg of beverage in orange juice or in the fed state, or one mid-low dose of the selected Arbaclofen Placarbil MR prototype tablet.
  Part 3 participants receive Regimens K and L in a randomised crossover manner as the first two treatments, followed by Regimens M and N in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A; Drug: Arbaclofen Placarbil MR Prototype B
- Part 3: Regimen M (Experimental): An optional regimen of one mid-low dose of the selected Arbaclofen Placarbil MR prototype tablet (if not previously dosed in Regimen L) or one mid-high dose of the selected Arbaclofen Placarbil MR prototype tablet taken under fasting conditions.
  Part 3 participants receive Regimens K and L in a randomised crossover manner as the first two treatments, followed by Regimens M and N in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A; Drug: Arbaclofen Placarbil MR Prototype B
- Part 3: Regimen N (Experimental): An optional regimen of one mid-high dose of the selected Arbaclofen Placarbil MR prototype tablet (if not previously dosed in Regimen M) or two mid-low dose of the selected Arbaclofen Placarbil MR prototype tablets.
  Part 3 participants receive Regimens K and L in a randomised crossover manner as the first two treatments, followed by Regimens M and N in a sequential manner.
  Interventions: Drug: Arbaclofen Placarbil MR Prototype A; Drug: Arbaclofen Placarbil MR Prototype B

INTERVENTIONS:
Drug: Arbaclofen Placarbil SR — One low dose oral tablet of Arbaclofen Placarbil sustained release (SR) in the fasted state.
  Arms: Part 1: Regimen C
Drug: Arbaclofen Placarbil MR Prototype A — One low dose oral tablet pf Arbaclofen Placarbil modified release (MR) Prototype A in the fasted state; this formulation may also be tested with 0.6 g/kg beverage diluted in orange juice
  Arms: Part 1: Regimen A; Part 1: Regimen D; Part 1: Regimen E; Part 2: Regimen F; Part 2: Regimen H; Part 2: Regimen I; Part 2: Regimen J; Part 3: Regimen K; Part 3: Regimen L; Part 3: Regimen M; Part 3: Regimen N
Drug: Arbaclofen Placarbil MR Prototype B — One low dose oral tablet of Arbaclofen Placarbil modified release (MR) Prototype B; this formulation may also be tested with 0.6 g/kg beverage diluted in orange juice
  Arms: Part 1: Regimen B; Part 1: Regimen D; Part 1: Regimen E; Part 2: Regimen F; Part 2: Regimen H; Part 2: Regimen I; Part 2: Regimen J; Part 3: Regimen K; Part 3: Regimen L; Part 3: Regimen M; Part 3: Regimen N
Drug: Arbaclofen Placarbil IR — One low dose oral capsule of Arbaclofen Placarbil immediate release (IR) in the fasted state.
  Arms: Part 2: Regimen G

SUMMARY:
Part 1

* To evaluate the pharmacokinetic (PK) profile of Arbaclofen Placarbil (AP) and R-baclofen following dosing of Arbaclofen Placarbil Modified Release (MR) Prototype A Tablet and Arbaclofen Placarbil MR Prototype B Tablet in healthy subjects
* To determine the relative bioavailability of AP and R-baclofen following dosing of Arbaclofen Placarbil MR Prototype A Tablet and Arbaclofen Placarbil MR Prototype B Tablet compared to the reference Arbaclofen Placarbil Sustained Release (SR) Tablets (low dose)
* To determine the relative bioavailability and PK of AP and R-baclofen following dosing of the selected MR prototype formulation(s) in the presence of beverage
* To provide additional information on the safety and tolerability of single doses of AP

Part 2

* To evaluate the PK profile of AP and R-baclofen following dosing of Arbaclofen Placarbil MR Prototype Tablets in healthy subjects
* To determine the relative bioavailability and PK of AP and R-baclofen following dosing of Arbaclofen Placarbil MR Prototype Tablets compared to the reference Arbaclofen Placarbil Immediate Release (IR) Capsule
* To provide additional information on the safety and tolerability of single doses of AP
* To determine the relative bioavailability and PK of AP and R-baclofen following dosing of a selected MR prototype formulation in the fed state (optional)
* To explore a possible in vitro in vivo correlation/relationship (IVIVC/IVIVR) for the Arbaclofen Placarbil MR Prototype Tablet Formulations

Part 3

* To determine the relative bioavailability of the selected Arbaclofen Placarbil MR Prototype Tablet in the presence of either beverage or food and/or
* To evaluate the PK profile (dose proportionality) of AP and R-baclofen following dosing of the selected Arbaclofen Placarbil MR Prototype A + B Tablet at different dose levels in healthy subjects
* To provide additional information on the safety and tolerability of single doses of AP

DETAILED DESCRIPTION:
For Parts 1, 2 and 3, participants will attend the clinical unit for a screening visit up to 28 days before dosing. For each treatment period, eligible subjects will be admitted to the clinical unit on the evening before dosing (Day -1). Participants will receive each regimen in the morning of Day 1 and will remain on site until 48 h post-dose. There will be a minimum washout period of 7 days between administration of each regimen. Where interim decisions occur, the interval between periods will be sufficient to permit the decision process.

Arbaclofen Placarbil MR Prototype Tablets will be administered in Part 1 and one prototype will be selected for development in Part 2 where the release rate of modified release (MR) prototype formulations will be optimised using a design space concept (at a fixed low dose).

A selected MR prototype formulation from Part 2 may be administered in Part 3 at up to 4 different dose levels (low, mid-low, mid-high, high). The suggested doses in Part 3 may be modified based on emerging safety and PK data from Part 2 of the study.

In Parts 2 and 3, there will be an option to dose selected Arbaclofen Placarbil MR Prototype Tablets in the fed state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Non-pregnant, non-lactating healthy females
* Body mass index of 18.0 to 30.0 kg/m^2 or, if outside the range, considered not clinically significant by the investigator
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent prior to any study-specific procedures
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the previous 3 months
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* Subjects who have previously been enrolled in this study
* History of any clinically significant drug/substance or alcohol abuse or disorders in the past 2 years
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Regular alcohol consumption <5 units per week on average
* Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and each admission
* Current smokers of e-cigarettes and nicotine replacement products and those who have smoked these products within the last 12 months
* Females of childbearing potential who are pregnant or lactating (female subjects must have a negative urine pregnancy test). A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle-stimulating hormone [FSH] concentration ≥40 IU/L)
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
* Clinically significant abnormal ECG as judged by the investigator, including a QT interval corrected using Fridericia's formula of >450 msec in males and >470 msec in females
* Positive drugs of abuse test result at screening and each admission (drugs of abuse tests are listed in the protocol)
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <70 mL/min using the Cockcroft-Gault equation
* History of cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease or psychiatric disorder, as judged by the investigator
* History of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system disorder (eg, Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system, or a history of significant head trauma within the past 2 years, or currently receiving anticonvulsant therapy for any reason
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol, hormone replacement therapy and hormonal contraceptives) or herbal remedies in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Part 1: Time to Maximum Concentration (Tmax) of Arbaclofen Placarbil (AP) and R-baclofen in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.

SECONDARY OUTCOMES:
Part 1: Maximum Observed Concentration (Cmax) of Arbaclofen Placarbil (AP) and R-baclofen in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: Concentrations at 12 Hours Post-dose (C12) of Arbaclofen Placarbil (AP) and R-baclofen in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose at 12 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: Concentrations at 24 Hours Post-dose (C24) of Arbaclofen Placarbil (AP) and R-baclofen in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose at 24 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: Area under the Concentration vs Time Curve From Time 0 to 12 Hours post-dose (AUC(0-12)) of Arbaclofen Placarbil (AP) and R-baclofen in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 12 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: Area under the Concentration vs Time Curve From Time 0 to 24 Hours post-dose (AUC(0-24)) of Arbaclofen Placarbil (AP) and R-baclofen in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 24 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: Area under the Concentration vs Time Curve From Time 0 to Last Measurable Concentration (AUC(0-last)) of Arbaclofen Placarbil (AP) and R-baclofen in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: Area under the Concentration vs Time Curve From Time 0 Extrapolated to Infinity (AUC(0-inf)) of Arbaclofen Placarbil (AP) and R-baclofen in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: Percentage of AUC(0-inf) Extrapolated Beyond Last Measured Time Point (AUC%extrap) of Arbaclofen Placarbil (AP) and R-baclofen in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: AP:R-baclofen AUC Ratios in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: AP:R-baclofen Cmax Ratios in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: The Slope of the Apparent Elimination Phase (lambda-z) in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: The Apparent Elimination Half-life (T1/2) in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: The Apparent Volume of Plasma Cleared of AP and R-baclofen per Unit Time Following Extravascular Dosing in Low Dose Arbaclofen Placarbil Modified Release (MR) Prototypes A + B | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in low dose arbaclofen placarbil modified release (MR) prototypes A and B.
Part 1: Relative Bioavailability of AP and R-baclofen following administration of Arbaclofen Placarbil Modified Release (MR) Prototypes A + B Compared to Reference Arbaclofen Placarbil Sustained Release (SR) | Day 1 (pre-dose), post-dose up to 48 hours
  The relative bioavailability of AP and R-baclofen following administration of arbaclofen placarbil modified release (MR) prototypes A + B compared to reference AP sustained release (SR), by calculation of Frel (relative bioavailability).
Part 1: Time to Maximum Concentration (Tmax) of AP and R-baclofen in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: Maximum Observed Concentration (Cmax) of AP and R-baclofen in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: Concentrations at 12 Hours Post-dose (C12) of AP and R-baclofen in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose at 12 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: Concentrations at 24 Hours Post-dose (C24) of AP and R-baclofen in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose at 24 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: Area under the Concentration vs Time Curve From Time 0 to 12 Hours post-dose (AUC(0-12)) of AP and R-baclofen in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 12 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: Area under the Concentration vs Time Curve From Time 0 to 24 Hours post-dose (AUC(0-24)) of AP and R-baclofen in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 24 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: Area under the Concentration vs Time Curve From Time 0 to Last Measurable Concentration (AUC(0-last)) of AP and R-baclofen in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: Area under the Concentration vs Time Curve From Time 0 Extrapolated to Infinity (AUC(0-inf)) of AP and R-baclofen in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: Percentage of AUC(0-inf) Extrapolated Beyond Last Measured Time Point (AUC%extrap) of AP and R-baclofen in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: AP:R-baclofen AUC Ratios in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: AP:R-baclofen Cmax Ratios in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: The Slope of the Apparent Elimination Phase (lambda-z) in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: The Apparent Elimination Half-life (T1/2) in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: The Apparent Volume of Plasma Cleared of AP and R-baclofen per Unit Time Following Extravascular Dosing in Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected MR prototype formulation(s) in the presence of beverage compared to when dosed with water only.
Part 1: Relative Bioavailability of AP and R-baclofen Following Administration of Selected MR Prototype Formulation(s) When Taken with Beverage Compared to Taken With Water | Day 1 (pre-dose), post-dose up to 48 hours
  Relative Bioavailability of AP and R-baclofen following administration of selected MR prototype formulation(s) when taken with beverage compared to taken with water, calculated by Frel.
Part 2: Time to Maximum Concentration (Tmax) of AP and R-baclofen in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low-dose MR prototype formulation(s).
Part 2: Maximum Observed Concentration (Cmax) of Arbaclofen Placarbil (AP) and R-baclofen in in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: Concentrations at 12 Hours Post-dose (C12) of Arbaclofen Placarbil (AP) and R-baclofen in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose at 12 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: Concentrations at 24 Hours Post-dose (C24) of Arbaclofen Placarbil (AP) and R-baclofen in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) Prototypes A + B | Day 1 (pre-dose), post-dose at 24 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: Area under the Concentration vs Time Curve From Time 0 to 12 Hours post-dose (AUC(0-12)) of Arbaclofen Placarbil (AP) and R-baclofen in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 12 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: Area under the Concentration vs Time Curve From Time 0 to 24 Hours post-dose (AUC(0-24)) of Arbaclofen Placarbil (AP) and R-baclofen in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 24 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: Area under the Concentration vs Time Curve From Time 0 to Last Measurable Concentration (AUC(0-last)) of Arbaclofen Placarbil (AP) and R-baclofen in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: Area under the Concentration vs Time Curve From Time 0 Extrapolated to Infinity (AUC(0-inf)) of Arbaclofen Placarbil (AP) and R-baclofen in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: Percentage of AUC(0-inf) Extrapolated Beyond Last Measured Time Point (AUC%extrap) of Arbaclofen Placarbil (AP) and R-baclofen in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: AP:R-baclofen AUC Ratios in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: AP:R-baclofen Cmax Ratios in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: The Slope of the Apparent Elimination Phase (lambda-z) in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: The Apparent Elimination Half-life (T1/2) in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: The Apparent Volume of Plasma Cleared of AP and R-baclofen per Unit Time Following Extravascular Dosing in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype(s) | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototypes.
Part 2: Relative Bioavailability of AP and R-baclofen following administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototypes Compared to Reference Arbaclofen Placarbil Immediate Release (IR) | Day 1 (pre-dose), post-dose up to 48 hours
  The relative bioavailability of AP and R-baclofen following administration of selected arbaclofen placarbil modified release (MR) Prototypes A + B compared to reference AP immediate release (IR), by calculation of Frel (relative bioavailability).
Part 2: Relative Bioavailability of AP and R-baclofen Following Administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  The relative bioavailability of AP and R-baclofen following administration of Arbaclofen Placarbil Modified Release (MR) Prototype in a fed state compared to a fasted state, by calculation of Frel (relative bioavailability).
Part 2: Time to Maximum Concentration (Tmax) of AP and R-baclofen Following Administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: Maximum Observed Concentration (Cmax) of AP and R-baclofen Following Administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: Concentrations at 12 Hours Post-dose (C12) of AP and R-baclofen Following Administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose at 12 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: Concentrations at 24 Hours Post-dose (C24) of AP and R-baclofen Following Administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose at 24 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: Area under the Concentration vs Time Curve From Time 0 to 12 Hours post-dose (AUC(0-12)) of AP and R-baclofen Following Administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 12 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: Area under the Concentration vs Time Curve From Time 0 to 24 Hours post-dose (AUC(0-24)) of AP and R-baclofen Following Administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 24 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: Area under the Concentration vs Time Curve From Time 0 to Last Measurable Concentration (AUC(0-last)) of AP and R-baclofen Following Administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: Area under the Concentration vs Time Curve From Time 0 Extrapolated to Infinity (AUC(0-inf)) of AP and R-baclofen Following Administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: Percentage of AUC(0-inf) Extrapolated Beyond Last Measured Time Point (AUC%extrap) of AP and R-baclofen Following Administration of Selected Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: AP:R-baclofen AUC Ratios in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  The relative bioavailability of AP and R-baclofen following administration of Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: AP:R-baclofen Cmax Ratios in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: The Slope of the Apparent Elimination Phase (lambda-z) in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: The Apparent Elimination Half-life (T1/2) in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 2: The Apparent Volume of Plasma Cleared of AP and R-baclofen per Unit Time Following Extravascular Dosing in Selected Low Dose Arbaclofen Placarbil Modified Release (MR) Prototype in Both a Fed and Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in selected low dose arbaclofen placarbil modified release (MR) prototype administered in a fed state compared to a fasted state.
Part 3: Relative Bioavailability of AP and R-baclofen in a Selected MR Prototype Formulation in the Fed State Compared to Fasted State | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. This outcome reports the relative bioavailability of AP and R-baclofen in a selected MR prototype formulation in the fed state compared to fasted, by calculation of Frel. An alternative is to compare the bioavailability of AP and R-baclofen when taken with beverage compared to taken with water, calculated by Frel.
Part 3: Time to Maximum Concentration (Tmax) of AP and R-baclofen in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: Maximum Observed Concentration (Cmax) of AP and R-baclofen in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: Concentrations at 12 Hours Post-dose (C12) of AP and R-baclofen in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose at 12 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: Concentrations at 24 Hours Post-dose (C24) of AP and R-baclofen in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose at 24 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: Area under the Concentration vs Time Curve From Time 0 to 12 Hours post-dose (AUC(0-12)) of AP and R-baclofen in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 12 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: Area under the Concentration vs Time Curve From Time 0 to 24 Hours post-dose (AUC(0-24)) of AP and R-baclofen in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 24 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: Area under the Concentration vs Time Curve From Time 0 to Last Measurable Concentration (AUC(0-last)) of AP and R-baclofen in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: Area under the Concentration vs Time Curve From Time 0 Extrapolated to Infinity (AUC(0-inf)) of AP and R-baclofen in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: Percentage of AUC(0-inf) Extrapolated Beyond Last Measured Time Point (AUC%extrap) of AP and R-baclofen in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: AP:R-baclofen AUC Ratios in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: AP:R-baclofen Cmax Ratios in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: The Slope of the Apparent Elimination Phase (lambda-z) in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: The Apparent Elimination Half-life (T1/2) in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Part 3: The Apparent Volume of Plasma Cleared of AP and R-baclofen per Unit Time Following Extravascular Dosing in a Selected MR Prototype Formulation at Different Dose Levels | Day 1 (pre-dose), post-dose up to 48 hours
  An optional outcome dependent upon decision-making in response to interim PK observations. Part of the pharmacokinetic profile of arbaclofen placarbil (AP) and R-baclofen in a selected MR prototype formulation at different dose levels.
Parts 1, 2 and 3: Participants with Adverse Events | Days 1-2 of each regimen
  The number of participants in categories of treatment-emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Global Director, Clinical Development, Study Director — Indivior Inc.
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No